CLINICAL TRIAL: NCT06338878
Title: PAtient Treatment Analysis: Hospital and Wide-ranging Out-of-hospital Care Assessment Yields Insights Into Heart Failure Outcomes
Acronym: PATHWAY-HF
Status: Recruiting | Type: Observational
Sponsor: Pr. Nicolas GIRERD (Other)
Responsible Party: Sponsor-Investigator, Pr. Nicolas GIRERD, Clinical Professor, Central Hospital, Nancy, France
Organization: Central Hospital, Nancy, France (Other)
Other Study IDs: 2023PI087
Record Dates: First submitted 2024-02-23; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a monocentric cohort study conducted in the cardiology department of Nancy hospital. The main purpose of the study is to document the global management strategy of patients hospitalized for heart failure and evaluate the association between patient's care and post-hospitalization outcome.

ELIGIBILITY:
Inclusion Criteria:

* Man or women ≥ 18 years
* Patients hospitalized for cardiac decompensation (ESC 2016 and 2021 criteria)

Exclusion Criteria:

* Patient expressing refusal to participate in research
* Patient who is a minor or under administrative protection
* Pregnant women
* Patient with ventricular assistance
* Patient with congenital heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for cardiac decompensation in the cardiology department of CHRU of Nancy,
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
All-cause post-hospitalization mortality | Within 1 year following hospital discharge
  Composite endpoint of all-cause post-hospitalization mortality and rehospitalization for heart failure with outcome 2
Rehospitalization for heart failure | Within 1 year following hospital discharge
  Composite endpoint of all-cause post-hospitalization mortality and rehospitalization for heart failure with outcome 1

SECONDARY OUTCOMES:
Percentage of maximum dose of each cardiotropic treatment indicated in heart failure according to ESC recommendations | Within 1 year following hospital discharge
Influenza and pneumococcal vaccination status | Within 1 year following hospital discharge
Evolution of renal function | During hospitalization for up to 2 months and within 1 year after discharge.
  Note: assessed by creatinine levels and GFR by CKD EPI
All-cause Rehospitalization | Within 1 year following hospital discharge
  Assessed by: Rehospitalization for any cause other than hear failure after discharge.
All-cause mortality | Within 1 year following hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas GIRERD, Study Chair — CHRU de Nancy; Olivier HUTTIN, Principal Investigator — CHRU de Nancy; Laura FILIPPETTI, Principal Investigator — CHRU de Nancy
Locations (1):
- CHRU de Nancy, Nancy, France